CLINICAL TRIAL: NCT01581918
Title: PHASE II STUDY TO EVALUATE EFFICACY AND SAFETY OF CARBAMAZEPINE FOR THE PREVENTION OF CHEMOTHERAPY-INDUCED NAUSEA AND VOMITING.
Brief Title: Efficacy and Safety Evaluation of Carbamazepine for Prevention of Chemotherapy-induced Nausea and Vomiting
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Faculdade de Medicina do ABC (Other)
Responsible Party: Principal Investigator, Felipe Melo Cruz, PHASE II STUDY TO EVALUATE EFFICACY AND SAFETY OF CARBAMAZEPINE FOR THE PREVENTION OF CHEMOTHERAPY-INDUCED NAUSEA AND VOMITING., Faculdade de Medicina do ABC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: thaiana123
Record Dates: First submitted 2012-04-19; First posted 2012-04-20 (Estimated); Last update posted 2012-04-24 (Estimated); Status verified 2012-04

CONDITIONS: Chemotherapy-induced Nausea and Vomiting
MeSH Terms: conditions — Vomiting | interventions — Carbamazepine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Carbamazepine — Patients will receive Carbamazepine in first chemotherapy cycle as planned: - One tablet (200mg) at night on third day before chemotherapy; - One tablet (200mg) every 12 hours on second day before chemotherapy; - One tablet (200mg) every 8 hours from the day before until fifth day after chemotherapy.

SUMMARY:
Nausea and vomiting are common problems for cancer patients. Half of them will experience these symptoms during the course of their disease, either because of the cancer itself or because of their treatment1. They are ranked by patients as two of the worst adverse effects of cancer chemotherapy and cause a negative impact on patient's functional, emotional, social and nutritional status and quality of life2,3.

Nowadays, a wide variety of antiemetic agents are available for the prevention and treatment of CINV. In this scenario, three classes play a critical role: Selective 5-HT3-receptor antagonists - approved for clinical practice in early 1990s, revolutionized the management of CINV representing the most effective agents in the treatment of acute emesis -, Corticosteroids - with unknown mechanism of action, effective when administered as single agents in patients receiving chemotherapy of low emetic potential but are most beneficial when used in combination with other antiemetic agents, potentiating their anti-emetic efficacy in both acute and delayed symptoms - and neurokinin 1 receptor antagonist - also effective against both acute and delayed emesis, but restricted utility in daily clinical practice because of its high cost.

DETAILED DESCRIPTION:
Meanwhile there are a lot of studies with these three classes of drugs, some efforts are being done to reach higher control rates of CINV with different drugs. In this scenario, in a randomized phase II placebo-controlled trial Cruz et. al. demonstrated that Gabapentin raises chemotherapy-induced nausea and vomiting control when associated with Dexametason and Ondasetron, suggesting that it could be a cost-effective alternative to neurokinin 1 receptor antagonists9, although, as we know, there aren't comparative studies with gabapentin and aprepitant. Guttuso et al demonstrated in an open clinical study the antiemetic effect of gabapentin in chemotherapy-induced acute (within 24hs) and delayed onset (days 2-5) nausea and vomiting in breast cancer patients with refractory emesis10.

Tan e cols showed higher complete and delayed nausea and vomiting control rates for olanzapine vs. aprepitant, in association with palonosetron and dexametason in highly and moderately emetogenic potential chemotherapy11. Navari e cols haven't found similar results although this comparison may not be done, since maintenance anti-emetic treatment was different between these studies12.

In a case report, Strohscheer I. & Borasio GD showed complete control of refractory nausea and vomiting in one patient with meningeal carcinomatosis treated with Carbamazepine13.

Carbamazepine is an available anticonvulsant largely used in Brazil. The aim of this study is to evaluate the role of Carbamazepine for the prevention of nausea and vomiting induced by moderate and highly emetogenic chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years old
* starting moderate or highly emetogenic chemotherapy defined as containing cisplatin,doxorrubicin or epirrubicin in higher doses than 60mg/m2, 50mg/m2 e 50mg/m2 respectively
* they must sign in the informed consent form.

Exclusion Criteria:

* previuos chemotherapy
* low emetogenic antiemetic potential
* disagree and don't sign in the consent form.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2011-12; Primary Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Efficacy of Carbamazepine | 120hours
  To evaluate complete protection (CP) of chemotherapy induced nausea and vomiting, defined as the percentage of patients without nausea or vomiting and the absence of use of rescue medication.

SECONDARY OUTCOMES:
Safety of Carbamazepine | 120hours
  Number of Adverse Events and possible impact in quality of life related to carbamazepine treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- ABC Medical School, Santo André, São Paulo, Brazil